CLINICAL TRIAL: NCT02317666
Title: Decreasing the Load? The Drug Burden Index - A Tool for Medication Reviews in Older People (the DBI TMO Study)
Brief Title: DBI - Tool for Medication Reviews in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Responsible Party: Principal Investigator, Katja Taxis, Professor of Pharmacotherapy and Clinical Pharmacy, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: the DBI TMO Study
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Polypharmacy; Cholinergic Antagonists
Keywords: polypharmacy; drug burden index; aged; medication review; cholinergic agents
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication Review (Experimental): Structured 5-step multidisciplinary medication review (STRIP method) performed by the pharmacist in collaboration with the general practitioner.
  Interventions: Procedure: Medication Review
- Delayed Medication Review (No Intervention): Patients in the control group will not undergo a medication review during the study period (delayed medication review).

INTERVENTIONS:
Procedure: Medication Review — A structured 5-step multidisciplinary medication review (STRIP method) as described in the multidisciplinary guidelines by the Nederlands Huisartsen Genootschap (2013) including the objective to reduce the DBI, performed by the pharmacist in collaboration with the general practitioner
  Arms: Medication Review

SUMMARY:
Older people often use medications with anticholinergic or sedative side effects which increase the risk of falling, fractures caused by falls and cognitive impairment. In the Netherlands, medication reviews are done by pharmacists in collaboration with the general practitioner to optimize medication use and reduce these adverse drug events. To maximize the benefits of medication reviews it is helpful to identify patients with high risk medication, yet few appropriate tools are available The Drug Burden Index (DBI) designed in Australia, calculates anticholinergic and sedative drug burden. This study evaluates whether the DBI can be used to identify patients with anticholinergic and sedative medication in need of a medication review. A clustered randomized controlled intervention study will be conducted. Per pharmacy (cluster), one pharmacist will perform the medication reviews. In each pharmacy, one half of eligible patients will be randomly allocated to the control group and the other half in the intervention group. Data will be collected at baseline and at follow-up, 3 months after the medication review has taken place. The study population includes community-dwelling patients aged ≥ 65, with polypharmacy (≥ 5 medications) and a DBI value ≥ 1 (n = 190) selected by 10 community pharmacists. The intervention consists of a structured 5-step multidisciplinary medication review (STRIP method) as described in the multidisciplinary guidelines of Dutch General Practitioners performed by the pharmacist in collaboration with the general practitioner. The main endpoint is the difference in proportion of patients having a decrease of the DBI ≥ 0.5 between the intervention and control group at 3 months follow up. Secondary outcomes are anticholinergic side effects, risk of falls, cognitive function, function of daily activity, hospital admission and mortality. All participants will be informed about the study and asked to provide informed consent. Data will be processed confidentially. Only the researcher will have access to the data. If required, the Dutch Inspection of Healthcare will also be granted access to the data for Inspection. The burden of patients will be kept at a minimum by trying to retrieve as much information as possible from patient's medical records and by using questionnaires and tests that were specifically developed for this population. In the investigators opinion, participation does not involve risks.

DETAILED DESCRIPTION:
Older people often use medications with anticholinergic or sedative side effects which increase the risk of falling, fractures caused by falls and cognitive impairment. In the Netherlands medication reviews are done by pharmacists in collaboration with the general practitioner to optimize the medication use and reduce these adverse drug events. To maximize the benefits of medication reviews it is helpful to identify patients with high risk medication, yet there are few tools to identify patients in need of a medication review. The Drug Burden Index (DBI) is a tool, designed in Australia, that calculates the burden of anticholinergic and sedative medications, taking into account a patient's dose. The DBI could be a useful tool to identify high risk patients who could benefit from medication reviews. The objective of this study is to evaluate whether the DBI can be used as a tool to identify patients with anticholinergic/sedative medication in need of a medication review. A single blinded clustered randomized controlled intervention study. Every pharmacy forms a cluster and per pharmacy one pharmacist will perform the medication reviews. In each pharmacy, one half of eligible patients will be randomly allocated to the control group and the other half in the intervention group. There are two measurements: at baseline and at follow-up, 3 months after the medication review has taken place. The study population includes community-dwelling patients aged ≥ 65, with polypharmacy (≥ 5 medications) and a DBI value ≥ 1 (n = 190) selected by 10 community pharmacists. The intervention consists a structured 5-step multidisciplinary medication review (STRIP method) as described in the multidisciplinary guidelines of the Dutch General Practitioners Society (Nederlands Huisartsen Genootschap, 2013) including the objective to reduce the DBI, performed by the pharmacist in collaboration with the general practitioner. The main endpoint is the difference in proportion of patients having a decrease of DBI ≥ 0.5 between the intervention and control group at follow up (3 months later). Secondary outcomes are the difference in proportion of patients having a DBI <1 between the intervention and control group at follow up (3 months later), the anticholinergic side effects, risk of falls, cognitive function, function of daily activity, hospital admission and mortality. All participants will be informed about the study. Informed consent will be asked from every participant. Data will be processed anonymously. Only the researcher will have access to the data. If required, the Dutch Inspection of Healthcare will also be granted access to the data for Inspection. The burden of patients will be kept at a minimum by trying to retrieve as much information as possible from patient's medical records and by using questionnaires and tests that were specifically developed for this population. In the investigators opinion, participation does not involve risks.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65,
* living independently,
* polypharmacy (≥ 5 medications),
* Drug Burden Index ≥ 1
* written informed consent

Exclusion Criteria:

* patients who have a limited life expectancy (<3 months)
* patients who urgently need a medication review and for whom postponing a medication review is unethical
* insufficient command of the Dutch language
* patients with advanced dementia.
* patients who received a medication review < 9 months before recruitment date

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 157 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
DBI decrease | 3 months
  The primary outcome is the difference in proportion of patients having a decrease of DBI ≥ 0.5 between the intervention and control group at follow-up.

SECONDARY OUTCOMES:
Anticholinergic side effects | 3 months
  Anticholinergic side effects, measured by the UKU side effect rating scale
Sedating side effects | 3 months
  Sedating side effects measured by a validated patient-reported adverse drug event questionnaire
Risk of falls | 3 months
  Risk of falls, measured by patients reports fall incidents and the "Up & Go" test to measure a patient's mobility
Cognitive Function | 3 months
  Cognitive function, measured by the Seven Minute Screen", the "Trailmaking Test A & B" and the "Digit Symbol Coding Test" of the Wechsler Adult Intelligence Scale III
Activities of Daily Living | 3 months
  Assessed with the Groningen Activities Restriction Scale [Dutch: Groningen Activiteiten Restrictie Schaal]
Quality of Life | 3 months
  as measured with the EQ-5D-3L
Hospitalisation | 3 months
  Incident hospital admission inferred from patients' medical records
Mortality | 3 months
  Incident mortality inferred from patients' medical records

CONTACTS AND LOCATIONS:
Overall Officials: Katja Taxis, PhD, Principal Investigator — University of Groningen
Locations (1):
- University of Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] van der Meer HG, Wouters H, Pont LG, Taxis K. Reducing the anticholinergic and sedative load in older patients on polypharmacy by pharmacist-led medication review: a randomised controlled trial. BMJ Open. 2018 Jul 19;8(7):e019042. doi: 10.1136/bmjopen-2017-019042. PMID 30030308
- [Derived] van der Meer HG, Wouters H, van Hulten R, Pras N, Taxis K. Decreasing the load? Is a Multidisciplinary Multistep Medication Review in older people an effective intervention to reduce a patient's Drug Burden Index? Protocol of a randomised controlled trial. BMJ Open. 2015 Dec 23;5(12):e009213. doi: 10.1136/bmjopen-2015-009213. PMID 26700279